CLINICAL TRIAL: NCT06052657
Title: Translation and Psychometric Properties of The Urdu Version of Identification of Functional Ankle Instability Questionnaire in Patients With Ankle Sprain
Brief Title: Urdu Version of Identification of Functional Ankle Instability Questionnaire
Status: Completed | Type: Observational
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Other Study IDs: REC-UOL-506-08-2023
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Ankle Sprains; Instability, Joint
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Functional instability should be considered as a potential cause of residual ankle impairment and instability. Even if neuromuscular anomalies are detected, the precise cause of injury and the most efficient prevention strategies remain uncertain. The use of standardized and validated research instruments is strongly advocated. This is due in part to the idea that it allows for international and cross-national comparison of results. Another assumption is that utilizing validated tools increases confidence that they are measuring what they are intended to measure. However, a previously validated tool does not guarantee its applicability in a new period, culture, or setting. The rationale of study is to provide a valid and reliable tool translated into native language of Urdu speaking populations so that self-evaluation of ankle instability can be assessed and re-assessed over the time. The questionnaire is translated into various languages including; French, Japanese, Brazilian, Persian, Thai, Malay, Greek, Chinese, Korean, Turkish and Spanish; whereas, Pakistani Urdu version has not yet studied. The present study fills this literature gap and serves a large proportion of Urdu community around the globe; specially, Pakistan. By measuring the psychometric properties of this scale in Urdu version, quantitatively strengthens up the evidence and patients themselves can report their exact level of disorder by answering a set of questions in their own language.

DETAILED DESCRIPTION:
Functional instability should be considered as a potential cause of residual ankle impairment and instability. Even if neuromuscular anomalies are detected, the precise cause of injury and the most efficient prevention strategies remain uncertain. The use of standardized and validated research instruments is strongly advocated. This is due in part to the idea that it allows for international and cross-national comparison of results. Another assumption is that utilizing validated tools increases confidence that they are measuring what they are intended to measure. However, a previously validated tool does not guarantee its applicability in a new period, culture, or setting. The rationale of study is to provide a valid and reliable tool translated into native language of Urdu speaking populations so that self-evaluation of ankle instability can be assessed and re-assessed over the time. The questionnaire is translated into various languages including; French, Japanese, Brazilian, Persian, Thai, Malay, Greek, Chinese, Korean, Turkish and Spanish; whereas, Pakistani Urdu version has not yet studied. The present study fills this literature gap and serves a large proportion of Urdu community around the globe; specially, Pakistan. By measuring the psychometric properties of this scale in Urdu version, quantitatively strengthens up the evidence and patients themselves can report their exact level of disorder by answering a set of questions in their own language.

For this purpose, the research conducted was a Cross-Sectional Validation Study involving 100 patients who had experienced ankle sprains. This study took place at the Department of Physical Therapy within the University of Lahore Teaching Hospital, situated on Defence Road in Lahore, spanning a nine-month duration following synopsis approval. The researchers employed a purposive sampling technique. Inclusion criteria encompassed individuals aged 18 and above, of both genders, diagnosed with ankle instability, and who had suffered from an ankle sprain for at least one month without receiving medical or physical therapy intervention during the study. Exclusions were made for participants displaying rheumatic or arthritic degenerative changes, those with a history of traumatic incidents like road accidents, individuals who had undergone lower extremity surgery, and participants with a current history of cancer. Ethical considerations were met as all participants provided written informed consent, and approval was obtained from the University of Lahore's Ethics Committee. Data collection involved using the translated Urdu version of Identification of Functional Ankle Instability Questionnaire Urdu Version (IDFAI-U).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were 18 years of age or older.
* Participants of both genders: male and female.
* Those diagnosed with ankle instability.
* Individuals who had experienced an ankle sprain for a minimum duration of one month.
* Participants who did not receive any medical treatment or physical therapy during the course of the study.

Exclusion Criteria:

* Participants who displayed rheumatic or arthritic degenerative changes.
* Those with a history of trauma, such as incidents from road traffic accidents.
* Individuals who had undergone surgery on their lower extremities.
* Participants who had an ongoing history of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ankle Sprain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Identification of functional ankle instability | 1 week
  Functional ankle instability (FAI) is the tendency of the foot to 'give way'. Identification of Functional Ankle Instability questionnaire (IdFAI) is a newly developed questionnaire to detect whether individuals meet the minimum criteria necessary for inclusion in an FAI population. IdFAI consists of 3 factors or domains: First factor focuses on the history of ankle sprain, second factor focuses on the initial ankle sprain, and the third factor focuses on the instability during ADL. Out of total 36 score, a score of 10 or lower indicates that the participant is unlikely to have FAI, whereas a total score of 11 or higher indicates that a participant is likely to have FAI.
Cumberland ankle instability tool | 1 week
  The Cumberland ankle instability tool (CAIT) is a 9-item scale measuring the severity of functional ankle instability. The total score of CAIT ranges from 0 to 30. Items focus on the degree of difficulty in performing different physical activities per ankle. The CAIT has the ability to discriminate between stable and unstable ankles and measures the severity of experienced functional instability, with a cut-off value of 27.5 points
Ankle Instability Instrument (AII) | 1 week
  The Ankle Instability Instrument (AII) was designed specifically to determine ankle instability. It captures the severity of the initial injury, history of ankle instability, and instability during activities of daily living (ADLs). It consists of 12 items related to the individual's perception of ankle instability and its impact on their daily life. Each item is scored on a 0 to 100 scale, with higher scores indicating less perceived instability and better ankle function.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrooj Hanif, MSPT MSK, Principal Investigator — University of Lahore; Hafiza Sana Ashraf, MSPT MSK, Study Director — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan